CLINICAL TRIAL: NCT04206163
Title: Somatostatin Receptor Imaging in Inflammatory Heart Disease
Brief Title: Somatostatin Receptor Imaging in Acute Myocarditis and Cardiac Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-001300-38
Record Dates: First submitted 2019-12-13; First posted 2019-12-20 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Acute Myocarditis; Cardiac Sarcoidosis
Keywords: Myocarditis; Cardiac sarcoidosis; Inflammatory cardiomyopathy; Cardiomyopathy; Heart disease; Cardiovascular disease; Somatostatin; 68Ga-DOTA-TOC; Positron emission tomography
MeSH Terms: conditions — Myocarditis; Cardiomyopathies; Heart Diseases; Cardiovascular Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acute myocarditis (Experimental): Included patients with clinically suspected acute myocarditis (n=30-40) will undergo a 68Ga-DOTA-TOC PET/CT and a blood sample will be taken. Furthermore, participants will undergo a contrast-enhanced MRI and endomyocardial biopsy (if clinically indicated) as part of the clinical routine work-up.
  Interventions: Diagnostic Test: 68Ga-DOTA-TOC PET/CT; Biological: Blood sample
- Cardiac sarcoidosis (Experimental): Included patients with clinically suspected cardiac sarcoidosis (n=30-40) will undergo a 68Ga-DOTA-TOC PET/CT and a blood sample will be taken. Furthermore, participants will undergo a contrast-enhanced MRI, 18F-FDG PET/CT and endomyocardial biopsy as part of the clinical routine work-up.
  Interventions: Diagnostic Test: 68Ga-DOTA-TOC PET/CT; Biological: Blood sample

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTA-TOC PET/CT — Somatostatin receptor imaging
Biological: Blood sample — Analysis of inflammatory biomarkers

SUMMARY:
This prospective imaging study investigates the diagnostic ability of Gallium-68 DOTA-TOC (68Ga-DOTA-TOC) positron emission tomography/computed tomography (PET/CT) in the clinical work-up of patients with 1) clinically suspected acute myocarditis (n=30-40) and 2) clinically suspected cardiac sarcoidosis (n=30-40) using clinical diagnostic criteria as well as endomyocardial biopsy as reference. Furthermore, 68Ga-DOTA-TOC PET/CT findings will be compared with results from contrast-enhanced magnetic resonance imaging (MRI) and in case of cardiac sarcoidosis even Fluorine-18 fluorodeoxyglucose (18F-FDG) PET/CT, which are both performed as part of the clinical routine work-up.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study
* Provision of written informed consent
* All patients between the age of 18 and 85 of both genders
* Newly clinically suspected acute myocarditis or newly clinically suspected cardiac sarcoidosis with or without known extra-cardiac sarcoid

Exclusion Criteria:

* Pregnancy or lactation
* Severe obesity (limited by the scanner)
* Other known significant cardiac disease, including previous myocarditis
* Known tumour disease, especially (neuro)endocrine tumours
* Terminal disease(s), advanced psychiatric disease and/or significant dementia
* Recent or current immunosuppressive treatment
* Recent or current somatostatin analogue (octreotide) therapy
* Known relative/absolute contraindications for contrast-enhanced MRI and/or PET/CT imaging
* Known contraindications for endomyocardial biopsy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-06-24 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Sensitivity of 68Ga-DOTA-TOC PET/CT versus contrast-enhanced MRI in patients with clinically suspected acute myocarditis (using clinical diagnostic criteria as well as endomyocardial biopsy as reference) | Completion of enrollment, approximately 2 years
Specificity of 68Ga-DOTA-TOC PET/CT versus contrast-enhanced MRI in patients with clinically suspected acute myocarditis (using clinical diagnostic criteria as well as endomyocardial biopsy as reference) | Completion of enrollment, approximately 2 years
Sensitivity of 68Ga-DOTA-TOC PET/CT versus contrast-enhanced MRI and 18F-FDG PET/CT in patients with clinically suspected cardiac sarcoidosis (using clinical diagnostic criteria as well as endomyocardial biopsy as reference) | Completion of enrollment, approximately 5 years
Specificity of 68Ga-DOTA-TOC PET/CT versus contrast-enhanced MRI and 18F-FDG PET/CT in patients with clinically suspected cardiac sarcoidosis (using clinical diagnostic criteria as well as endomyocardial biopsy as reference) | Completion of enrollment, approximately 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian L Polte, MD, PhD, MSc, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No